CLINICAL TRIAL: NCT04916314
Title: Testing the Effectiveness of a Low Carbohydrate Diet With Remote Support for Patients With Type 2 Diabetes in Primary Care, on Weight and Glycaemic Control: a Randomised Controlled Trial
Brief Title: REmote SUpport for Low-Carbohydrate Treatment of Type 2 Diabetes
Acronym: RESULT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15434
Record Dates: First submitted 2021-05-26; First posted 2021-06-07 (Actual); Results first posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-02

CONDITIONS: Type 2 Diabetes Mellitus in Obese
Keywords: Diet; Low-Carbohydrate; Digital Intervention
MeSH Terms: interventions — Diet, Carbohydrate-Restricted

STUDY DESIGN:
Masking Description: The nature of the intervention means it is not possible to mask providers or patients
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Carbohydrate Diet (Experimental): . The intervention involves diet, activity and behaviour change components. It comprises a three-month remote behavioural change programme with mentoring from a registered dietitian or nutritionist (health coach), peer group support, structured education articles and activity tracking technology. These elements are accessed via a smartphone or web-based application. Each participant will also receive a hard copy of an instructional handbook and a recipe book.
  Interventions: Behavioral: Low Carbohydrate diet
- Standard NHS type 2 diabetes care (No Intervention): Participants randomised to the control group will receive no additional intervention, and will continue to receive their usual NHS diabetes care from their general practice.

INTERVENTIONS:
Behavioral: Low Carbohydrate diet — The intervention is a three-month remote behavioural change programme with mentoring from a registered dietitian or nutritionist (health coach), encouraging adoption of a low energy, low-carbohydrate diet, peer group support, structured education articles and activity tracking technology. These elements are accessed via a smartphone or web-based application; each participant additionally receives an instructional handbook, and recipe book (+/-wireless weighing and activity tracking technology).
  Arms: Low Carbohydrate Diet

SUMMARY:
Excess adiposity is a key causal factor in developing type 2 diabetes and weight loss improves glycaemia and can put diabetes in to remission. There is evidence that low carbohydrate diets also reduce glycaemia. The aim of this trial is to test a behavioural support programme delivered remotely to reduce energy intake and carbohydrate intake in particular to improve glycaemic control in people recently diagnosed with type 2 diabetes. We will recruit participants from general practice diabetes registers who were diagnosed within the past six years and who want to and are able to follow an app-based behavioural support programme to change their diet and have a BMI of at least 27kg/m2 (≥30kg/m2 if of white European ethnicity). They will be individually randomised 1:1 using simple randomisation to either intervention or a no-intervention control. Blinding of participants or their clinicians is impossible. The intervention comprises a 12-week behavioural support programme delivered by app or web, which provides group-based peer support, recipes for food providing low energy meals that are low in carbohydrate. The programme is delivered by a commercial company who run NHS commissioned programmes in several areas of the UK. Clinicians will adjust medication for hypertension and diabetes as needed. The co-primary outcomes are change in participants' HbA1c from baseline to 3 months and baseline to 1 year, with p-value adjustment to reflect multiple testing. The secondary outcomes are remission from diabetes, weight change, change in cardiovascular risk factors, and change in quality of life at 3 months and 1 year. The trial will assess whether this app-based programme improves outcomes for people with type 2 diabetes relative to usual care.

DETAILED DESCRIPTION:
This is an individually randomised controlled trial. Participants, recruited via GP practices, will be randomised 1:1 with simple randomisation and no stratification to either the intervention group or control (usual care). They will be enrolled in the study for 1 year, of which the intervention (dietary support via the app) will run for 3 months. Most study procedures will be conducted online or remotely (by telephone) including: screening, eligibility assessment, informed consent, randomisation, engagement with the app-based intervention. Participants will be asked to attend 3 face to face appointments for the research study at their local GP practice for measurements to be taken (weight, blood pressure) and blood tests, at baseline, 3 months and 1 year, and will have 1 additional telephone contact with their GP or practice nurse before starting the intervention. Face to face appointments will be incorporated with routine clinical appointments when possible.

The investigators aim to recruit 100 participants via their GP practices. Based on a conservative response rate of 10% from similar previous studies, the investigators will approach approximately 1000 eligible individuals from approximately 10 GP practices in England. The primary care provider will search their electronic registers for eligible individuals and GPs will screen out those to whom it would be inappropriate to send a letter inviting them to enrol and referring them to a website to give informed consent.

Once consent has been given, participants will click on a link to the electronic data capture system database which will be activated following their consent, to complete the baseline assessment. All participants will complete a 2 part baseline assessment, firstly online and then at their GP practice.

1. Online:

   Participants will be asked to complete a baseline questionnaire requesting demographic information and their current medication, and the standard questionnaires that will be used in the study (the Problem Areas in Diabetes (PAID) score, the EQ5D (quality of life assessment), and a 24 hour dietary recall questionnaire ("Intake24 dietary assessment tool", where participants are asked to record all food and drink intake in the last 24 hours). This will also further assess whether people are sufficiently able to complete online trial procedures, and only those who complete the questionnaire will be randomised. Participants will be informed in the Participant Information Sheet that they will only be able to enter the study after completing the questionnaire fully in one attempt as the system will not allow them to go back into the questionnaire to answer the remaining questions later. This should take less than 30 minutes to complete.
2. At the GP practice (visit 1) Having completed the online assessment, participants will be asked (via message on their screen on completing the assessment, and followed up via email) to book the in-person portions of their baseline assessment at their GP practice for measures which cannot be conducted online. At this appointment, their height, weight and blood pressure will be measured and recorded, and a blood sample taken for baseline values (HbA1c, lipid profile, liver function tests).

The clinician will randomise the participant at the baseline appointment. This is an individually randomised 1:1 to 2 arms: Intervention (12 week, app-based dietary support), or control (usual care; no active additional intervention). The randomisation will be conducted using the in-built randomisation software. This ensures full allocation concealment as information on future allocations is not accessible to the person randomising. Due to the nature of the intervention it will not be possible to blind members of the study team or participants to allocation.

Participants randomised to the intervention group will receive an email giving 12 weeks of access to the app/website. The intervention involves diet, activity and behaviour change components. It comprises a three-month remote behavioural change programme with mentoring from a registered dietitian or nutritionist (health coach), peer group support, structured education articles and activity tracking technology. These elements are accessed via a smartphone or web-based application. Each participant will also receive a hard copy of an instructional handbook and a recipe book.

Participants randomised to the intervention group will consult their GP to adjust medication as appropriate to avoid hypotension or hypoglycaemia following a guideline.

Participants randomised to the control group will receive no additional intervention, and will continue to receive their usual NHS diabetes care from their general practice.

All Participants will be followed up after 3 months (visit 2) and at 12 months (visit 3). At this appointment they will have the same procedures as at their baseline assessment repeated: their weight and blood pressure will be recorded, and blood tests taken (3 sample tubes - for HbA1c, lipid profile and liver function). Participants will be asked to complete the same online questionnaires (PAID score, EQ5D, and 24 hour dietary recall) as they completed at baseline, and serious adverse events and events of concern (serious hypoglycaemia) will be recorded.

A purposively sampled proportion of participants from the intervention group (aiming to achieve diversity of age, race, and success and engagement with the programme measured by weight/HbA1c outcomes and engagement metrics respectively) will be contacted via telephone for a semi-structured interview to discuss their experience of the intervention, after they complete the 3 month intervention period. Interviews will last approximately 30 minutes. With participants consent this will be audio-recorded.

The duration of the SAE recording period for each participant lasts from their enrolment on to the study, to their completion of the study.

The study results will be reported in accordance with the CONSORT (Consolidated Standards of Reporting Trials) 2010 statements. A full analysis plan will be prepared and finalised before any data analysis.

The primary statistical analysis of efficacy outcomes will be carried out on the basis of intention-to-treat (ITT). This is, after randomisation, participants will be analysed according to their allocated intervention group irrespective of what intervention they actually receive. The investigators will endeavour to obtain full follow-up data on every participant to allow full ITT analysis, but the investigators will inevitably experience the problem of missing data due to withdrawal, loss to follow up, or non-response to questionnaire items.

The investigators will analyse the primary continuous outcome with a linear model adjusting for baseline value of the relevant variable where relevant. For exploratory analyses, the investigators will use analogous models, but interpret the data in an exploratory manner rather than confirmatory. For binary outcomes (e.g. remission), the investigators will test for a difference in proportions using logistic regression.

Based on previous studies of this intervention(5) and studies in similar populations(3), an 8-10mmol/mol change in HbA1c at 12 months in the intervention group in those who engage with the programme (SD 8.6mmol/mol), with a 1-2mmol/mol (SD 6mmol/mol) change in the control group is estimated. With α and β set at 0.05 this would require approximately 48 participants; however to power for a co-primary outcome would require 72 to 88 participants in total (allowing for variability in estimated effect size). In similar trials of behavioural interventions an expected retention to follow up of >80%; allowing for the online nature of this trial, and the retention rates of observational studies of this intervention the investigators will aim to recruit 100 participants to allow for cumulative attrition at the intervention sign-up, engagement, and follow up stages. The results from the trial will be prepared as comparative summary statistics (difference in proportions or means) with 95% confidence intervals. All the tests will be done at a 5% two-sided significance level.

This study is funded by the Wellcome Trust (220551/Z/20/Z) and the NIHR Oxford Biomedical Research Centre.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Male or Female, aged 40 years or above.
* Diagnosed with current type 2 diabetes (i.e. not in remission) in the last 6 years
* BMI of ≥27kg/m2 (≥30kg/m2 if ethnicity recorded as white)
* Has a smartphone or computer with internet access (and the correct operating system requirements to use the intervention programme)
* Are able to complete the eligibility and baseline assessments online
* Would like to make changes to their diet or lifestyle to improve their diabetes control, lose weight, or improve their general health

Exclusion Criteria:

* Unable to understand the study materials and interventions
* Currently following a weight loss programme (defined as a structured, prescribed and monitored programme and not a self-directed weight loss attempt)
* Pregnant, breastfeeding, or planning to become pregnant during the course of the study
* History of bariatric surgery, including gastric banding
* Currently using insulin therapy
* Proliferative diabetic retinopathy, or maculopathy.
* Recent myocardial infarction or stroke (<3 months)
* Renal failure (chronic kidney disease stage 4 or 5)
* Current active treatment for cancer (other than skin cancer treated with curative intent by local treatment only)
* Their doctor does not feel they are appropriate to participate for another reason (e.g. active eating disorder diagnosis, significant psychological disturbance)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Aveyard, FRCP, Principal Investigator — University of Oxford
Locations (1):
- University of Oxford, Warwick, Select A Region, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
IPD will be available upon direct request to the study team
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will be available indefinitely when the investigators have completed their analysis, about 1 year after final follow-up.
Access Criteria: Request is for bona fide reasons from an organisation whose mission is to benefit the public good.

REFERENCES:
- [Derived] Morris E, Scragg J, Stevens R, Albury C, Aveyard P, Jebb SA. A randomised controlled trial of a low-carbohydrate digitally-supported weight loss programme for type 2 diabetes. NPJ Digit Med. 2025 Dec 2;8(1):739. doi: 10.1038/s41746-025-02116-w. PMID 41331050

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Low Carbohydrate Diet | Standard NHS Type 2 Diabetes Care
Started | 55 | 60
Completed | 52 | 59
Not Completed | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Low Carbohydrate Diet: The intervention involves diet, activity and behaviour change components. It comprises a three-month remote behavioural change programme with mentoring from a registered dietitian or nutritionist (health coach), peer group support, structured education articles and activity tracking technology. These elements are accessed via a smartphone or web-based application. Each participant will also receive a hard copy of an instructional handbook and a recipe book.
- Total: Total of all reporting groups
Arm/Group | Low Carbohydrate Diet | Standard NHS Type 2 Diabetes Care | Total
Number analyzed (Participants) | 55 | 60 | 115
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.1 (9.6) | 57.3 (8.8) | 58.7 (9.2)
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 51 | 58 | 109
  Asian | 3 | 1 | 4
  Black, mixed or other ethnicity | 1 | 1 | 2
HbA1c [Mean (Standard Deviation); unit: mmol/mol] | 51.3 (10.2) | 57.4 (12.9) | 54.5 (12.0)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 31 | 32 | 63
  Male | 23 | 27 | 50
  Prefer not to say | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Participants' HbA1c
Description: Change in participants' HbA1c from baseline to 3 months
Time Frame: Baseline to 3 months
Measure: Mean (Standard Deviation); unit: mmol/mol
Arm/Group | Low Carbohydrate Diet | Standard NHS Type 2 Diabetes Care
Number analyzed (Participants) | 55 | 60
mmol/mol | -2.3 (7.9) | -2.4 (8.5)
Statistical Analysis 1: Comparison: Low Carbohydrate Diet vs Standard NHS Type 2 Diabetes Care; Test type: Superiority; p = 0.8, Mixed Models Analysis — Omnibus likelihood ratio test for significant change in co-primary outcomes at 3 or 12 months; Mean Difference (Net) = -0.7, 95% CI 2-sided [-5 to 3.6]

2. Primary Outcome: Change From Baseline in Participants' HbA1c
Description: Change in participants' HbA1c from baseline to 12 months
Time Frame: Baseline to 12 months
Measure: Mean (Standard Deviation); unit: mmol/mol
Arm/Group | Low Carbohydrate Diet | Standard NHS Type 2 Diabetes Care
Number analyzed (Participants) | 55 | 60
mmol/mol | 0.4 (11.9) | -1 (15.8)
Statistical Analysis 1: Comparison: Low Carbohydrate Diet vs Standard NHS Type 2 Diabetes Care; Test type: Superiority; p = 0.8, Mixed Models Analysis — omnibus likelihood ratio test for significant change in co-primary outcomes at 3 or 12 months; Mean Difference (Net) = -1.5, 95% CI 2-sided [-5.7 to 2.8]

3. Secondary Outcome: Diabetes Remission at 12 Months
Description: Number of participants meeting consensus definition for remission from type 2 diabetes at 1 year
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Low Carbohydrate Diet | Standard NHS Type 2 Diabetes Care
Number analyzed (Participants) | 55 | 60
Participants | 4 | 1

4. Secondary Outcome: Weight Change From Baseline
Description: Change in participants' weight from baseline to 3 and 12 months
Time Frame: 3 months,1 year
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Low Carbohydrate Diet | Standard NHS Type 2 Diabetes Care
Number analyzed (Participants) | 55 | 60
kg
  Weight change from baseline at 3 months | -3.6 (3.6) | -0.7 (5.9)
  Weight change from baseline at 12 months | -2.4 (5.3) | -2.7 (5.9)

5. Secondary Outcome: Change in Systolic Blood Pressure, From Baseline
Description: Change in participants' systolic blood pressure from baseline
Time Frame: 3 months, 1 year
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Low Carbohydrate Diet | Standard NHS Type 2 Diabetes Care
Number analyzed (Participants) | 55 | 60
mmHg
  Systolic BP change from baseline to 3 months | -2.1 (12.3) | -2.9 (13)
  Systolic BP change from baseline to 12 months | -1.6 (14.2) | -0.9 (15.2)

6. Secondary Outcome: Change in Diastolic Blood Pressure, From Baseline
Description: Change in participants' diastolic blood pressure from baseline to 3 and 12 months
Time Frame: 3 months, 1 year
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Low Carbohydrate Diet | Standard NHS Type 2 Diabetes Care
Number analyzed (Participants) | 55 | 60
mmHg
  Diastolic BP change from baseline to 3 months | -2.1 (9.1) | -3.2 (8)
  Diastolic BP change from baseline to 12 months | -0.21 (0.61) | -0.35 (0.98)

7. Secondary Outcome: Change in LDL Cholesterol From Baseline
Description: Change in participants' LDL cholesterol from baseline to 3 and 12 months
Time Frame: 3 months, 1 year
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Low Carbohydrate Diet | Standard NHS Type 2 Diabetes Care
Number analyzed (Participants) | 55 | 60
mmol/L
  LDL cholesterol change from baseline to 3 months | -0.04 (0.52) | -0.10 (0.49)
  LDL cholesterol change from baseline to 12 months | -0.22 (0.62) | 0.04 (0.15)

8. Secondary Outcome: Change in Total Cholesterol:HDL Ratio From Baseline
Description: Change in participants' total cholesterol:HDL ratio from baseline to 3 and 12 months
Time Frame: 3 months, 1 year
Measure: Mean (Standard Deviation); unit: (ratio; no units)
Arm/Group | Low Carbohydrate Diet | Standard NHS Type 2 Diabetes Care
Number analyzed (Participants) | 55 | 60
(ratio; no units)
  Total cholesterol:HDL ratio change from baseline to 3 months | -0.11 (0.71) | -0.36 (0.87)
  Total cholesterol:HDL ratio change from baseline to 12 months | -0.35 (0.67) | -0.55 (1.09)

9. Secondary Outcome: Change in HDL Cholesterol, From Baseline
Description: Change in participants' HDL cholesterol from baseline to 3 and 12 months
Time Frame: 3 months, 1 year
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Low Carbohydrate Diet | Standard NHS Type 2 Diabetes Care
Number analyzed (Participants) | 55 | 60
mmol/L
  HDL cholesterol change from baseline to 3 months | 0.03 (0.17) | 0.04 (0.15)
  HDL cholesterol change from baseline to 12 months | 0.07 (0.39) | 0.04 (0.15)

10. Secondary Outcome: Change in Triglycerides, From Baseline
Description: Change in participants' triglycerides from baseline to 3 and 12 months
Time Frame: 3 months, 1 year
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Low Carbohydrate Diet | Standard NHS Type 2 Diabetes Care
Number analyzed (Participants) | 55 | 60
mmol/L
  Triglycerides change from baseline to 3 months | -0.07 (1.03) | -0.29 (1.28)
  Triglycerides change from baseline to 12 months | -0.25 (0.86) | -0.19 (1.29)

11. Secondary Outcome: Change in ALT From Baseline
Description: Change in participants' ALT from baseline to 3 and 12 months
Time Frame: 3 months, 1 year
Measure: Mean (Standard Deviation); unit: iU/L
Arm/Group | Low Carbohydrate Diet | Standard NHS Type 2 Diabetes Care
Number analyzed (Participants) | 55 | 60
iU/L
  Change in ALT from baseline to 3 months | -3.3 (13) | -2.4 (10.9)
  Change in ALT from baseline to 12 months | -2.1 (15.4) | -4.1 (16.6)

12. Secondary Outcome: Change in Diabetes Related Quality of Life and Distresses - Problem Areas In Diabetes (PAID) Score From Baseline
Description: Change in participants' PAID score from baseline to 3 and 12 months. (Minimum- maximum score; 0-100). Lower score indicating lower diabetes burden.
Time Frame: 3 months, 1 year
Measure: Mean (Standard Deviation); unit: numerical score
Arm/Group | Low Carbohydrate Diet | Standard NHS Type 2 Diabetes Care
Number analyzed (Participants) | 55 | 60
numerical score
  Change in PAID score from baseline to 3 months | -12.3 (18.1) | -11.4 (16.2)
  Change in PAID score from baseline to 12 months | -14.8 (17.2) | -10 (16.5)

13. Secondary Outcome: Change in Participants' EQ5D Score From Baseline
Description: Change in participants' EQ5D score from baseline to 3 and 12 months. (Score minimum-maximum is 0-1, VAS is 0-100).
Time Frame: 3 months, 1 year
Measure: Mean (Standard Deviation); unit: numerical score
Arm/Group | Low Carbohydrate Diet | Standard NHS Type 2 Diabetes Care
Number analyzed (Participants) | 55 | 60
numerical score
  Change in EQ5D-5L index value from baseline to 3 months | 0.059 (0.135) | 0.0004 (0.149)
  Change in EQ5D-5L index value from baseline to 12 months | 0.041 (0.152) | 0.001 (0.014)
  Change in EQ5D-5L VAS score from baseline to 3 months | 5.2 (17.6) | 4.0 (19.7)
  Change in EQ5D-5L VAS score from baseline to 12 months | 4.5 (12.2) | 5.9 (22.4)

14. Other Pre Specified Outcome: Dietary Intake Patterns
Description: Data will be collected on change in dietary intake patterns (via Intake24 24 hour dietary recall questionnaire)
Time Frame: Baseline, 3 months, 1 year
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Engagement With Programme; 'Learn' Component of the Programme
Description: Data will be collected on measures of engagement with one of the three main components of the programme ("Learn") via the app programme
Time Frame: Baseline, 3 months, 1 year
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Engagement With Programme; 'Track' Component of the Programme
Description: Data will be collected on measures of engagement with one of the three main components of the programme ("Track") via the app programme
Time Frame: Baseline, 3 months, 1 year
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Engagement With Programme; 'Support' Component of the Programme
Description: Data will be collected on measures of engagement with one of the three main components of the programme ("Support"), via the app programme
Time Frame: Baseline, 3 months, 1 year
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Participants' Experience of Using the App-based Support
Description: Interviews with participants
Time Frame: 3 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 year
Description: There were no events deemed serious and related to the study procedures
Arm/Group | Low Carbohydrate Diet | Standard NHS Type 2 Diabetes Care
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/60
Other Adverse Events (participants affected / at risk) | 1/55 | 10/60
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Carbohydrate Diet (N=55) | Standard NHS Type 2 Diabetes Care (N=60)
Unplanned hospital admission (Investigations) | 1 (1) | 10 (10) — Unplanned hospital admissions - not for elective or planned procedures

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-16): https://cdn.clinicaltrials.gov/large-docs/14/NCT04916314/Prot_SAP_000.pdf